CLINICAL TRIAL: NCT04881006
Title: A Single-Dose, Bioequivalence, Pivotal Study of Two Formulations of Dapagliflozin 10 mg Tablets Under Fed Conditions
Brief Title: Bioequivalence of Dapagliflozin 10 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2020-4926
Record Dates: First submitted 2021-04-30; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): Manufactured by Jiangsu Hansoh Pharmaceutical Group Co., Ltd. Drug: Dapagliflozin 10 mg tablets A single 10 mg dose (1 tablet) of the assigned drug product will be administered according to the randomization scheme with 240±5 mL of room temperature potable water.
  Interventions: Drug: Dapagliflozin 10 mg tablets
- Reference Product (Active Comparator): Manufactured by AstraZeneca Pharmaceuticals LP Drug: Farxiga® 10 mg tablets A single 10 mg dose (1 tablet) of the assigned drug product will be administered according to the randomization scheme with 240±5 mL of room temperature potable water.
  Interventions: Drug: Farxiga® 10 mg tablets

INTERVENTIONS:
Drug: Dapagliflozin 10 mg tablets — Manufactured by Jiangsu Hansoh Pharmaceutical Group Co., Ltd.
  Arms: Test Product
Drug: Farxiga® 10 mg tablets — Manufactured by AstraZeneca Pharmaceuticals LP
  Arms: Reference Product

SUMMARY:
The primary objective of this study is to evaluate the bioequivalence between:

* Dapagliflozin 10 mg tablets from Jiangsu Hansoh Pharmaceutical Group Co., Ltd.,China; and
* Farxiga® 10 mg tablets from AstraZeneca Pharmaceuticals LP, USA; after a single-dose in healthy subjects under fed conditions. The secondary objective of this study is to evaluate the safety and tolerability of the study treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking, male and female subjects, 18 years of age or older.
2. BMI ≥19 and ≤30 kg/m2.
3. Females may be of childbearing or non-childbearing potential:

   * Childbearing potential:

     o Physically capable of becoming pregnant
   * Non-childbearing potential:

     * Surgically sterile (i.e., both ovaries removed, uterus removed, or bilateral tubal ligation); and/or
     * Postmenopausal (no menstrual period for at least 12 consecutive months without any other medical cause).
4. Willing to use acceptable, effective methods of contraception.
5. Able to tolerate venipuncture.
6. Be informed of the nature of the study and give written consent prior to any study procedure.

Exclusion Criteria:

1. Known history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Known or suspected carcinoma.
3. Known history or presence of hypersensitivity or idiosyncratic reaction to dapagliflozin or any other drug substances with similar activity.
4. Known history or presence of congestive heart failure, volume depletion, hypotension, and/or electrolyte imbalances.
5. Known history or presence of pancreatitis, DM, lactic acidosis, or acute or chronic metabolic acidosis, including diabetic ketoacidosis.
6. Known history or presence of clinically significant angioedema.
7. Known history or presence of clinically significant lactose, galactose, or fructose intolerance.
8. Presence of hepatic or renal dysfunction.
9. History of malabsorption within the last year or presence of clinically significant gastrointestinal disease.
10. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
11. Known history or presence of genital mycotic infections.
12. History or presence of Fournier's gangrene (necrotising fasciitis of the perineum).
13. History of drug or alcohol addiction requiring treatment.
14. Presence of urinary tract infection, urosepsis, or pyelonephritis.
15. Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
16. Positive test result for urine drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, phencyclidine, and tricyclic antidepressants) or urine cotinine.
17. Difficulty fasting or consuming high-fat or standard meals.
18. Use of tobacco or nicotine-containing products within 6 months prior to drug administration.
19. Females who:

    * Have discontinued or changed the use of implanted, intrauterine, intravaginal, or injected hormonal contraceptives within 6 months prior to drug administration;
    * Have discontinued or changed the use of oral or patch hormonal contraceptives within 1 month prior to drug administration;
    * Are pregnant (serum hCG consistent with pregnancy); or
    * Are lactating.
20. Donation or loss of whole blood (including clinical trials):

    * ≥50 mL and <500 mL within 30 days prior to drug administration;
    * ≥500 mL within 56 days prior to drug administration.
21. Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
22. On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw food diet).
23. Have had a tattoo or body piercing within 30 days prior to drug administration.
24. Have clinically significant findings in vital signs measurements.
25. Have clinically significant findings in a 12-lead ECG.
26. Have clinically significant abnormal laboratory values.
27. Have significant diseases.
28. Have clinically significant findings from a physical examination.
29. Use of any of the following within 30 days prior to drug administration:

    * Drugs that alter gastrointestinal pH/movement (e.g., omeprazole, ranitidine);
    * Enzyme-modifying drugs known to induce/inhibit hepatic drug metabolism;
    * Diuretics (e.g., thiazide and loop diuretics);
    * Insulin and insulin secretagogues (e.g., sulphonyl ureas);
    * Mefenamic acid;
    * Pioglitazone;
    * Rifampin;
    * Simvastatin; or
    * Valsartan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Cmax | up to Day 10 post-administration
  Peak plasma concentration (Cmax) of Dapagliflozin in plasma after administration of the test and the reference products. In Period 1 and Period 2, blood samples were collected at prior to dosing (0-hour) and 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, and 48 hours after drug administration.
AUCt | up to Day 10 post-administration
  The area under the plasma concentration-time curve from zero to last measurable concentration (AUCt) of Dapagliflozin in plasma after administration of the test and the reference products. In Period 1 and Period 2, blood samples were collected at prior to dosing (0-hour) and 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, and 48 hours after drug administration.
AUCinf | up to Day 10 post-administration
  The area under the plasma concentration-time curve from zero to infinity (AUCinf) of Dapagliflozin in plasma after administration of the test and the reference products. In Period 1 and Period 2, blood samples were collected at prior to dosing (0-hour) and 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.33, 3.67, 4, 4.5, 5, 6, 8, 12, 16, 24, 36, and 48 hours after drug administration.

SECONDARY OUTCOMES:
Adverse Events | up to Day 10 post-administration.
  AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with the treatment. All AEs are classified according to version 23.1 of MedDRA and reported with respect to incidence, frequency, severity, duration, relationship to the investigational medicinal product, action taken, and outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharma Medica Research Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No